CLINICAL TRIAL: NCT05321862
Title: Exploratory Study Evaluating the Relevance of [68Ga]Ga-PentixaFor for Initial Staging and Detection of Minimal Residual Disease in Multiple Myeloma Patients Eligible for Autologous Stem Cell Transplantation Less Than 66 Years Included in the Prospective IFM 2020-02.
Brief Title: Relevance Evaluation of [68Ga]Ga-PentixaFor for Initial Staging and Detection of Minimal Residual Disease in Multiple Myeloma Patients.
Acronym: PENTI-MIDAS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: MIDAS inclusions terminated before first inclusion in PENTI-MIDAS
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC22_0150
Record Dates: First submitted 2022-03-24; First posted 2022-04-11 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-PentixaFor (Experimental)
  Interventions: Drug: [68Ga]Ga-PentixaFor

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — Tomography by Emission of Positons (PET) with the radiopharmaceutic [68Ga]Ga-PentixaFor

SUMMARY:
The aim of our study is to confirm the relevance of PET using [68Ga]Ga-PentixaFor ligand, in comparison with FDG, for initial staging and detection of minimal residual disease in multiple myeloma patients eligible for autologous stem cell transplantation less than 66 years.

The prognostic value of positive CXCR4 expression will also be assessed and [68Ga]Ga-PentixaFor/FDG discordances explored.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are identical to inclusion criteria in MIDAS study (EudraCT Number: 2020-005216-21, ClinicalTrials.gov Identifier: NCT04934475) .

Exclusion Criteria:

* Non inclusion criteria are identical to non inclusion criteria in MIDAS study (EudraCT Number: 2020-005216-21, ClinicalTrials.gov Identifier: NCT04934475) added with:

  1. eGFR < 50 ml/min by MDRD or CKDEPI.
  2. Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years.
  3. Patient with uncontrolled insulin-dependent or non-insulin-dependent diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 6 months
  To determine the sensitivity of [68Ga]Ga-PentixaFor-PET to detect Multiple Myeloma lesions [Bone marrow (BM) lesions and/or extra-medullary disease (EMD)] at the time of initial diagnosis in high risk MM patients included in the MIDAS study.

SECONDARY OUTCOMES:
Specificity, positive predictive value (PPV) and negative predictive value (NPV) of [68Ga]Ga-PentixaFor-PET. | 1 month
  The specificity (PPV and NPV) of [68Ga]Ga-PentixaFor-PET at the time of initial diagnosis will be assessed by patient and lesion analysis using the same definitions of TP and FN as for the primary objective.
Prognostic impact of FDG-PET and of [68Ga]Ga-PentixaFor-PET depending on the uptake detected by each imaging technique. | 1 month
  The prognostic impact of FDG-PET and [68Ga]Ga-PentixaFor-PET based on the number of lesions detected of uptake by each imaging technique will be evaluated by assessing the impact of these data on the PFS and OS. PFS is defined as the time from the start of treatment to relapse or progression. OS is defined as the time from the start of first treatment to death.
Discrepancies rate between FDG-PET and [68Ga]Ga-PentixaFor-PET and factors associated with. | 1 month and 6 months
  * We will consider as discordant a lesion positive by FDG-PET but negative by [68Ga]Ga-PentixaFor-PET and/or a lesion negative by FDG-PET but positive by [68Ga]Ga-PentixaFor-PET.
Correlation between FDG-PET and [68Ga]Ga-PentixaFor-PET uptakes evaluated by SUV. | 1 month
  [68Ga]Ga-PentixaFor and FDG uptakes assessed by SUV.
Correlation between FDG-PET and [68Ga]Ga-PentixaFor-PET uptakes evaluated by the RNAseq data evaluated on the myelogram. | 1 month
  [68Ga]Ga-PentixaFor and FDG uptakes assessed by the quantitative expression of biological markers on myelogram (including expression of the gene coding for hexokinases).
Prognostic impact of FDG-PET and [68Ga]Ga-PentixaFor-PET depending on the positivity, number and intensity of uptake detected by each imaging technique. | 6 months
  The prognostic impact of [68Ga]Ga-PentixaFor-PET after therapy will be determined by evaluating the impact of a decrease uptake and/or a normalization of images on PFS and OS.
Link between FDG-PET, [68Ga]Ga-PentixaFor-PET results and minimal residual disease evaluated by NGS. | 6 months
  FDG-PET, [68Ga]Ga-PentixaFor-PET results (positive/negative) and minimal residual disease evaluated by NGS (positive/negative).
Tolerance of [68Ga]Ga-PentixaFor-PET. | 1 month and 6 months
  Tolerance of [68Ga]Ga-PentixaFor will be assessed by clinical monitoring of the patient for 1 hour after [68Ga]Ga-PentixaFor injection. Clinical data will be collected prior and 5/10 min after [68Ga]Ga-PentixaFor injection before acquisition (at 60 min after the injection) and at the end of acquisition (at approximately 80 min after the injection).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided